CLINICAL TRIAL: NCT05227599
Title: BRAVE: Building Resilience and Values Through E-health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-55183
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Survivorship

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily Diary Method Cohort (Other): Participants will be asked to complete a self-report questionnaire that has been validated to assess daily affect. There are 5 items assessing positive affect (joyful, cheerful, happy, lively, proud) and 5 items assessing negative affect (miserable, mad, afraid, scared sad). The respondent is asked to rate these 10 different feelings on a 5-point Likert scale from 1, "not much or not at all" to 5, "a lot."
  Interventions: Other: Online survey questionnaire

INTERVENTIONS:
Other: Online survey questionnaire — Participants will complete a brief online survey every morning and evening within 1 hour of waking and 1 hour of going to sleep. The surveys will be a combination of measures used to assess affect, stress, and symptoms

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of tracking survivors' and their caregivers, stressors, affect, and symptoms using an electronic diary method, in the time period surrounding their routine check- up with their oncologist.

ELIGIBILITY:
Inclusion Criteria:

1. 11-25 years old
2. previously received a pediatric cancer diagnosis and treatment for such
3. completed cancer treatment <5 years ago, in remission
4. Own a smart phone or tablet
5. are English proficient

Exclusion Criteria:

* no cognitive, motor, or sensory deficits that could preclude completion of study measures.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Online survey questionnaire | 21 days
  participants will complete a brief online survey every morning and evening within 1 hour of waking and 1 hour of going to sleep

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Mueller, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, San Francisco, California, United States